CLINICAL TRIAL: NCT02964624
Title: Response of Osteoarthritis Biomarkers After a Rehabilitation Program
Brief Title: Ostearthritis Biomarkers and Rehabilitation
Acronym: Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Ohio State University (Other); Federal University of São Paulo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Osteoarthritis
Record Dates: First submitted 2016-10-21; First posted 2016-11-16 (Estimated); Last update posted 2023-09-22 (Actual); Status verified 2018-07

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; biomarkers; HMGB1; knee
MeSH Terms: conditions — Osteoarthritis | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rehabilitation (Other): The rehabilitation protocol will consist of three exercise session/week for eight weeks
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — Protocol will consist of three exercise/week for eight weeks. Each session will begin with the evaluation of pain by the volunteer. Starting with a warm up exercise in a cycle ergometer (CEE), for 5 minutes at free cadence, then the intensity will be set at 90% of the intensity obtained during the incremental test and maintained for 10 min. Afterward, four sets of three different resistance exercises (RE) will be performed at 70% of the load correspondent to 1RM test with one minute interval between sets and exercises. During CEE Borg scale will be taken every two minutes and during RE the OMNI scale taken at the end of every set to monitor the intensity. At the end of the session, cool down global stretching exercises for inferior members will be performed and the VAS evaluated.

SUMMARY:
Osteoarthritis (OA) is the most common type of degenerative joint disease. Furthermore, despite its incidence being amongst the highest in chronic diseases, effective biomarkers, diagnostic aids and imaging technology are not available to assist in the management of OA. Mounting evidence suggests that non-pharmacological treatment such as exercise/physical therapy may lower the risk for onset or progression of OA by mitigating inflammation. However, the mechanical unloading and overloading, as seen in disuse and overuse, lead to upregulation of several proinflammatory molecules and enhance tissue degradation, whereas, dynamic moderate mechanical loading exerts anti-inflammatory and anti-catabolic effects on articular cartilage by suppressing mediators of inflammation. However, the lack of robust biomarkers to measure the effectiveness of physical therapies, represent a critical gap in biotechnology, obliterating the progress in the optimal application of these therapies. Our central hypothesis is that the circulating levels of specific molecules could serve as robust biomarkers for quantitative measures of OA burden, prognosis, progression or treatment efficacy. The objective of this project is to identify and evaluate mediators that serve as biomarkers of OA progression and treatment. Recently, high mobility group box chromosomal protein 1 (HMGB-1) has been suggested to be markedly upregulated in OA. However, presently there are no inhibitors of HMGB1 that could be used therapeutically. Previous results showed that that gentle exercise is the only tool that can mitigate HMGB1 production by local and systemic macrophages, and thus inflammation. Serum concentration of HMGB1 will be evaluate as a biomarker in OA patients and relate it to the functional capacity of knee joints in OA patients after rehabilitation protocol (RP). The RP will consist of three rehabilitation session/week during eight weeks. The efficacy of a RP will be evaluated by functional scale Western Ontario & McMaster Universities Osteoarthritis (WOMAC), Scale for the measurement of health related quality of life using EuroQol five dimensions questionnaire (EuroQOL), Visual Analog Scale (VAS), and physical function tests. Besides all clinical assessment, serum levels of classical pro-inflammatory cytokines, hyaluronan and HMGB1 will be evaluated. A correlation of physical improvement after RP and serum biomarkers will be performed.

DETAILED DESCRIPTION:
Detailed Description:

Methods/Design

1. Participants after being textually and verbally informed about their rights, benefits and possible risks, objectives and methodologies of this study, all participants will sign a free and informed consent form.
2. Study Design Prior to the rehabilitation protocol (RP), participants will perform one adaptation session to all the functional tests that will be applied to minimize learning bias. In the second session after 5 minutes warm up in a cycle ergometer (CEE), the Time Up and Go (TUG) test will be applied, followed by the isometric strength test. In the third day, after the same warm up, one repetition maximum testing will be conducted. At the end of the RP, all the tests will be repeated. Blood samples will be collected at baseline (day 0), 1 month (day 30 after RP) and at 2 months (day 60 after RP).

2.1. Rehabilitation protocol (RP) The RP will consist of 3 exercise session/week for 8 weeks. Each session will begin with the evaluation of pain by the participants. If the pain is higher than four, an analgesic protocol (AP) containing ultra-sound, laser or transcutaneous electrical nerve stimulation (TENS) will be applied. After the AP, the participant will just execute the rehabilitation protocol if the pain decreased to or lower than four. Starting with a warm up exercise in a cycle ergometer (CEE), for 5 minutes at free cadence, then the intensity will be set at 90% of the intensity obtained during the incremental test (see item 2.2a) and maintained for 10 min. Afterward, four sets (8-12 repetitions) of three different resistance exercises (RE) (leg press, knee extension and knee flexion) will be performed at 70% of the load correspondent to 1RM test (see item 2.2b) with one minute interval between sets and exercises. During CEE Borg scale will be taken every two minutes and during RE the omnibus (OMNI) scale taken at the end of every set to monitor the intensity. At the end of the session, cool down global stretching exercises for inferior members will be performed and the VAS evaluated again. Ten seconds of tension for each stretching position targeting the hamstrings, quadriceps, gluteus maxim ums, gastrocnemius, thigh adductors and abductors.

2.2. Rehabilitation intensity parameters.

1. Cycle ergometer incremental test (CEEIT). After 5 minutes warm up at free cadence in a cycle ergometer, the intensity will be increased every 3 minutes until the participants register 11 to 13 in Borg scale which is consider a moderate intensity and to be correlated to blood lactate concentration threshold and anaerobic threshold, respectively .
2. One repetition maximum. The test starts with a warm up of 5 to 10 repetitions with estimated moderate load (± 40-60% of 1RM). After 1 minute rest 3 to 5 repetitions are performed with higher load (±60-80% of 1RM) with 5 minutes rest. Then one attempt at estimated 1RM is given. If the participants fail to lift the load for two repetitions the test stops, otherwise after 5 minutes rest the load is increased and the test is performed again. Only five attempts per day are permitted to maintain the test reliable.

Sample size calculation The estimation of sample size was determined on the basis of a greater improvement of subscale physical function of the WOMAC score, using G.Power 3.15 software. Based on 10% expected difference between baseline measure and after RP and a standard deviation of 30 on physical function of WOMAC, 65 participants are needed with significance level of 0.05, and power of 80%.

ELIGIBILITY:
Inclusion Criteria:

* Women and men aged 45-65 years
* Clinical knee osteoarthritis according to the American College of Rheumatology Clinical Criteria
* Kellgren and Lawrence (KL) radiographic osteoarthritis grade 2 and 3 (mild to moderate radiographic osteoarthritis)

Exclusion Criteria:

* Severe knee osteoarthritis according to the KL classification (grade 4)
* Other known major musculoskeletal impairments in the lower extremities or the back or prostheses in any joint of the lower extremities
* Known serious coronary heart diseases or cancer
* Body mass index >35
* Scheduled for surgery in any joint
* Persons who already perform sports related moderate physical activity more than two times a week
* History of knee replacement surgery or high tibial osteotomy;
* Any knee surgery or corticosteroid injections within the previous 6 months;
* Miss more than two rehabilitation sessions during the program or more than two consecutive sessions.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline to month 2 in Western Ontario and McMasters Universities Osteoarthritis (WOMAC) Index score | Baseline and 2 month
  Participants will answer the questionnaire WOMAC for the assessment of lower extremity pain, stiffness and physical function during daily activities. The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). For each item, the possible range of scores is therefore 0-100. Items are summed for each subscale, resulting in possible ranges as follows: pain=0-500, stiffness=0-200, physical function=0-1700. Most commonly, a total WOMAC score is created by summing the items for all three subscales. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations. The collected data will be present through study completion, an average of 1 year.

SECONDARY OUTCOMES:
Change from baseline to month 2 in TUG test | Baseline and 2 month
  The purpose of TUG is to test basic mobility skills of frail elderly persons. The test consists of the time measurement in seconds for a participant to rise from sitting from a standard arm chair, walk 3 meters, turn, walk back to the chair, and sit down. The unity of measure is time in seconds. It will also be performed on day 0 (baseline) and day 60 (2 months after RP). The collected data will be present through study completion, an average of 1 year.
Change from baseline to month 2 in VAS analysis. | Baseline and 2 month
  The pain VAS is a unidimensional measure of pain intensity, which has been widely used in diverse adult populations, including those with rheumatic diseases. The unity of measures is in points. It will also be performed on day 0 (baseline) and day 60 (2 months after RP). The collected data will be present through study completion, an average of 1 year.
Change from baseline in proinflammatory cytokines and biomarkers of cartilage breakdown in blood | Baseline, 1 month and 2 month after RP
  Serum samples will be obtained by venous blood collection (3 vacutainer tubes, each containing 6 mL). The venous blood will be collected from the antecubital vein on day 0 (baseline), day 30 (1 month after RP) and day 60 (2 months after RP). After being centrifuged at 1800 g for 10 minutes, samples will be stored at -80 degrees Celsius in 1 mL aliquots. Serum concentrations of cytokines (Interleukin (IL)-6, IL-8, IL-1β, IL-10, IL-17, and tumor necrosis factor (TNF)-alpha) will be simultaneously evaluated. Serum HMGB1 and serum cartilage oligomeric matrix protein (COMP), will be analyzed by specific kits. The unity of measure is ng/mL. The collected data will be present through study completion, an average of 1 year.
Change from baseline to month 2 in Health-related quality of life (EuroQOL-5D, EQ-5D) | Baseline and 2 month
  Health-related QOL will be assessed by the EQ-5D. The unity of measure is in points. Also, day 0 (pre-RP) and day 60 (after 2 months of RP) will be evaluated for assessment. The collected data will be present through study completion, an average of 1 year.
Change from baseline to month 2 in Radiographic knee osteoarthritis progression (joint space and KL score) | Baseline and 2 month
  Radiological examination of conventional radiographic procedure will be performed at baseline and at day 60 after RP (2 month) for assessment. The degree of osteoarthritis can vary 0 to 5. The collected data will be present through study completion, an average of 1 year.
Change from baseline to month 2 in Isometric strength testing | Baseline and 2 month
  Isometric strength will be measured by the peak torque (PT) obtained during knee extension (PTE) and flexion (PTF) maximal voluntary contraction (MVC) using an isokinetic dynamometer (Biodex, Shirley, NY). During test the participants was seated and securely strapped the dynamometer chair. For knee extension MVC the thigh and leg angle will be 75° (0° = total extension) and for knee flexion MVC thigh-leg angle will be 40° (0° = total extension). Two attempts of five seconds MVC will be performed for each joint movement, with 3 minutes of interval between them. The unity of measure is Newtons per meter (N.m). The isometric PTE and PTF will be determined as the highest PT values between attempts. It will also be performed on day 0 (pre-RP) and day 60 (after 2 months of RP) for assessment. The data will be present through study completion, an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Ferretti, PhD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (2):
- Brazil (2):
  - Universidade Federal de Sao Paulo, São Paulo, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Weinstein SL, Jacobs JJ, Goldberg MJ. Osteoarthritis of the knee. N Engl J Med. 2006 Jun 8;354(23):2508-9; author reply 2508-9. doi: 10.1056/NEJMc060815. No abstract available. PMID 16760456
- [Background] Kapoor M, Martel-Pelletier J, Lajeunesse D, Pelletier JP, Fahmi H. Role of proinflammatory cytokines in the pathophysiology of osteoarthritis. Nat Rev Rheumatol. 2011 Jan;7(1):33-42. doi: 10.1038/nrrheum.2010.196. Epub 2010 Nov 30. PMID 21119608
- [Background] Cross M, Smith E, Hoy D, Nolte S, Ackerman I, Fransen M, Bridgett L, Williams S, Guillemin F, Hill CL, Laslett LL, Jones G, Cicuttini F, Osborne R, Vos T, Buchbinder R, Woolf A, March L. The global burden of hip and knee osteoarthritis: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1323-30. doi: 10.1136/annrheumdis-2013-204763. Epub 2014 Feb 19. PMID 24553908
- [Background] McAlindon TE, Bannuru RR, Sullivan MC, Arden NK, Berenbaum F, Bierma-Zeinstra SM, Hawker GA, Henrotin Y, Hunter DJ, Kawaguchi H, Kwoh K, Lohmander S, Rannou F, Roos EM, Underwood M. OARSI guidelines for the non-surgical management of knee osteoarthritis. Osteoarthritis Cartilage. 2014 Mar;22(3):363-88. doi: 10.1016/j.joca.2014.01.003. Epub 2014 Jan 24. PMID 24462672
- [Background] Zhang W, Moskowitz RW, Nuki G, Abramson S, Altman RD, Arden N, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis, Part II: OARSI evidence-based, expert consensus guidelines. Osteoarthritis Cartilage. 2008 Feb;16(2):137-62. doi: 10.1016/j.joca.2007.12.013. PMID 18279766
- [Background] Altman R, Asch E, Bloch D, Bole G, Borenstein D, Brandt K, Christy W, Cooke TD, Greenwald R, Hochberg M, et al. Development of criteria for the classification and reporting of osteoarthritis. Classification of osteoarthritis of the knee. Diagnostic and Therapeutic Criteria Committee of the American Rheumatism Association. Arthritis Rheum. 1986 Aug;29(8):1039-49. doi: 10.1002/art.1780290816. PMID 3741515
- [Background] Hsueh MF, Onnerfjord P, Kraus VB. Biomarkers and proteomic analysis of osteoarthritis. Matrix Biol. 2014 Oct;39:56-66. doi: 10.1016/j.matbio.2014.08.012. Epub 2014 Aug 30. PMID 25179675
- [Background] Kraus VB, Blanco FJ, Englund M, Henrotin Y, Lohmander LS, Losina E, Onnerfjord P, Persiani S. OARSI Clinical Trials Recommendations: Soluble biomarker assessments in clinical trials in osteoarthritis. Osteoarthritis Cartilage. 2015 May;23(5):686-97. doi: 10.1016/j.joca.2015.03.002. PMID 25952342
- [Background] Terada C, Yoshida A, Nasu Y, Mori S, Tomono Y, Tanaka M, Takahashi HK, Nishibori M, Ozaki T, Nishida K. Gene expression and localization of high-mobility group box chromosomal protein-1 (HMGB-1)in human osteoarthritic cartilage. Acta Med Okayama. 2011 Dec;65(6):369-77. doi: 10.18926/AMO/47262. PMID 22189477
- [Background] Hunt MA, Pollock CL, Kraus VB, Saxne T, Peters S, Huebner JL, Sayre EC, Cibere J. Relationships amongst osteoarthritis biomarkers, dynamic knee joint load, and exercise: results from a randomized controlled pilot study. BMC Musculoskelet Disord. 2013 Mar 27;14:115. doi: 10.1186/1471-2474-14-115. PMID 23530976
- [Background] Andersson U, Harris HE. The role of HMGB1 in the pathogenesis of rheumatic disease. Biochim Biophys Acta. 2010 Jan-Feb;1799(1-2):141-8. doi: 10.1016/j.bbagrm.2009.11.003. PMID 20123076
- [Background] Imamura M, Ezquerro F, Marcon Alfieri F, Vilas Boas L, Tozetto-Mendoza TR, Chen J, Ozcakar L, Arendt-Nielsen L, Rizzo Battistella L. Serum levels of proinflammatory cytokines in painful knee osteoarthritis and sensitization. Int J Inflam. 2015;2015:329792. doi: 10.1155/2015/329792. Epub 2015 Mar 2. PMID 25821631
- [Background] Li ZC, Cheng GQ, Hu KZ, Li MQ, Zang WP, Dong YQ, Wang WL, Liu ZD. Correlation of synovial fluid HMGB-1 levels with radiographic severity of knee osteoarthritis. Clin Invest Med. 2011 Oct 1;34(5):E298. doi: 10.25011/cim.v34i5.15673. PMID 21968272
- [Derived] Campedelli RR, Jardim MRS, Antonioli E, de Oliveira FBD, Agarwal S, Ferretti M. Effect of simplified exercise program on quality of life, biomarkers, pain and muscle strength of individuals with knee osteoarthritis. Einstein (Sao Paulo). 2025 Dec 1;23:eAO1192. doi: 10.31744/einstein_journal/2025AO1192. eCollection 2025. PMID 41379149